CLINICAL TRIAL: NCT03609801
Title: A Randomized Trial of the Duluth Model and ACTV for Domestic Violence
Brief Title: The Duluth Model and ACTV for Domestic Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Amie Zarling, Associate Professor, Iowa State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-007
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Domestic Violence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACTV (Experimental): Achieving Change Through Values-Based Behavior (ACTV) - pronounced "ACTIVE" - is a new Batterers Intervention Program (BIP) for domestic violence offenders. ACTV was developed as a collaboration between researchers, practitioners, and the criminal justice system in the state of Iowa (Zarling, Lawrence, Oregno, 2017). It is based on Acceptance and Commitment Therapy (ACT; Hayes, Strosahl, & Wilson, 1999), which is an evidence-based cognitive-behavioral psychotherapy. ACTV is an innovative BIP in two primary ways; first, ACTV applies the ACT model to the treatment of domestic violence, and second, ACTV is specifically designed for use in the correctional setting as part of criminal justice programming.
  Interventions: Behavioral: ACTV
- The Duluth Model (Active Comparator): The Duluth Model Men's Nonviolence Classes is the most widely used BIP. The Duluth Model is based on the premise that domestic abuse happens when men believe they have the right to authority over women who are their intimate partners. The Duluth Model's Men's Nonviolence Classes (The Duluth Model for short) help men stop battering and explore the consequences of the violence for themselves, their partner and their children.
  Interventions: Behavioral: The Duluth Model

INTERVENTIONS:
Behavioral: ACTV — Achieving Change Through Values-Based Behavior (ACTV) - pronounced "ACTIVE" - is a new intervention program for domestic violence offenders. ACTV was developed as a collaboration between researchers, practitioners, and the criminal justice system in the state of Iowa (Zarling, Lawrence, Oregno, 2017). It is based on Acceptance and Commitment Therapy (ACT; Hayes, Strosahl, & Wilson, 1999), which is an evidence-based cognitive-behavioral psychotherapy. ACTV is innovative in two primary ways; first, ACTV applies the ACT model to the treatment of domestic violence, and second, ACTV is specifically designed for use in the correctional setting as part of criminal justice programming.
  Arms: ACTV
Behavioral: The Duluth Model — The Duluth Model is based on the premise that domestic abuse happens when men believe they have the right to authority over women who are their intimate partners. The Duluth Model Men's Nonviolence Classes help men stop battering and explore the consequences of the violence for themselves, their partner and their children.
  Arms: The Duluth Model

SUMMARY:
The purpose of this research is to compare the effectiveness of two interventions for intimate partner violence (IPV). In most states, men who are convicted of domestic assault court-mandated to complete a Batterers Intervention Program (BIP) as part of their sentencing. The most commonly used BIP is based on The Duluth Model, which has been shown to decrease the recidivism of IPV offenders, but only marginally. The Duluth Model is a group intervention based on feminist theory and cognitive behavioral therapy. A new BIP called Achieving Change Through Values-Based Behavior (ACTV) has recently been developed by the PI as an alternative to Duluth. ACTV is currently being used statewide within the Department of Corrections (DOC) in Iowa. ACTV is a group intervention that utilizes acceptance and mindfulness techniques in addition to techniques from cognitive behavior therapy. The current study will use a randomized control trial to compare Duluth and ACTV, in order to assess the interventions' relative impact reducing IPV behaviors (physical aggression, psychological aggression, stalking, harassment, etc). Data on these outcomes will be collected via official criminal justice reports (i.e., criminal charges) as well as reports from victims. Other processes and outcomes of interest (attitudes toward women, emotion regulation, parenting behaviors, etc) will be collected from offenders.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* First time domestic assault offender
* Domestic assault must be against an intimate partner
* Must be on supervision/probation

Exclusion Criteria:

* Participation in any previous ACT-based or Duluth Model programming

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 799 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Domestic assault recidivism | One year time period following BIP
  Domestic assault charges (per criminal justice data)
Conflict Tactics Scale | Start and end of BIP, then one year later
  Psychological (subscale min-max= 0-48), physical (subscale min-max= 0-72), and sexual (subscale min-max= 0-42) aggression (per victim reports); higher values = greater frequency of aggressive acts

SECONDARY OUTCOMES:
Acceptance and Action Questionnaire-II (AAQ-II) | Start and end of BIP
  Experiential avoidance (per offender self-report); min-max = 7-49; higher scores = greater experiential avoidance
Male Role Norms Inventory-Revised | Start and end of BIP
  Sexist beliefs and attitudes; min-max = 21-147; higher scores = greater agreement with traditional gender roles and sexist beliefs

CONTACTS AND LOCATIONS:
Overall Officials: Amie Zarling, Ph.D., Principal Investigator — Iowa State University
Locations (1):
- 5th Judicial District Department of Corrections, Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zarling A, Berta M, Weems CF. Changes in Sexist Beliefs and Psychological Flexibility Among Men Court-Mandated to Domestic Violence Programs. J Interpers Violence. 2025 Sep 24:8862605251368854. doi: 10.1177/08862605251368854. Online ahead of print. PMID 40990942
- [Derived] Zarling A, Russell D. A randomized clinical trial of acceptance and commitment therapy and the Duluth Model classes for men court-mandated to a domestic violence program. J Consult Clin Psychol. 2022 Apr;90(4):326-338. doi: 10.1037/ccp0000722. PMID 35446078